CLINICAL TRIAL: NCT02047162
Title: Randomized, Double-blind, Placebo-controlled Trial of the Impact of Bismuth Subsalicylate on Antimicrobial Use Among Adult Diarrhea Outpatients in Pakistan
Brief Title: Impact of Bismuth Subsalicylate on Antimicrobial Use Among Adult Diarrhea Outpatients--Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Procter and Gamble (Industry); Health Oriented Preventive Education (Other)
Responsible Party: Principal Investigator, Anna Bowen, Medical Epidemiologist, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 6469
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Diarrhea
Keywords: diarrhea; gastroenteritis; antimicrobial drug resistance; antimicrobial agents; Pakistan; ambulatory care; bismuth
MeSH Terms: conditions — Diarrhea; Gastroenteritis | interventions — bismuth subsalicylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bismuth subsalicylate (Experimental): Bismuth subsalicylate, 262 mg/chewable tablet, 2 tablets every hour as needed up to 16 tablets per 24 hours, for up to 48 hours.
  Interventions: Drug: Bismuth subsalicylate
- Placebo (Placebo Comparator): Placebo chewable tablets, 2 every hour as needed up to 16 tablets per 24 h, for up to 48 h.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bismuth subsalicylate
  Other Names: Pepto-Bismol
  Arms: Bismuth subsalicylate
Other: Placebo — Chewable tablets identical to intervention tablets, but missing the bismuth subsalicylate
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn whether bismuth subsalicylate can reduce use of antibiotics among adults with diarrhea in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 15 - 65 years old
* Presenting with mild to moderate, non-bloody, acute diarrhea (≥3 loose stools/day for <3 days) to participating health care settings
* For whom the study physicians recommend antimicrobial treatment

Exclusion Criteria:

* Is pregnant
* Requires hospitalization
* Has signs or symptoms of septicemia
* Has a primary complaint of another acute illness
* Has a serious chronic illness
* Has an allergy to aspirin
* Has been exposed to antimicrobial or antidiarrheal medications within 72 hours of enrollment
* Previously enrolled in study

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
use of antimicrobial medications | within 5 days of enrollment

SECONDARY OUTCOMES:
Patient's perceived need for antibiotics | Within 48 h of enrollment
additional care obtained for diarrhea | within 48 h of enrollment
  Use of antidiarrheal medications, visits to other health professionals for diarrhea or complications of diarrhea, or expenditures on consultations and treatments for diarrheal illness
Additional care obtained for diarrheal illness | within 5 days of enrollment
  Use of antidiarrheal medications, visits to other health professionals for diarrhea or complications of diarrhea, or expenditures on consultations and treatments for diarrheal illness
Disease severity and duration | within 5 days of enrollment
  Time to first formed stool Number of stools during first 48 h of observation Duration of abdominal pain Duration of nausea Time to resolution of illness (any of the following symptoms: diarrhea, nausea, vomiting, abdominal pain) Severity of all symptoms of illness
Patient experience with the study drug | within 5 days of enrollment
  i. Satisfaction with resolution of symptoms ii. Satisfaction with esthetics of study medication iii. Adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bowen, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- HOPE, Karachi, Pakistan

REFERENCES:
- [Derived] Bowen A, Agboatwalla M, Pitz A, Salahuddin S, Brum J, Plikaytis B. Effect of Bismuth Subsalicylate vs Placebo on Use of Antibiotics Among Adult Outpatients With Diarrhea in Pakistan: A Randomized Clinical Trial. JAMA Netw Open. 2019 Aug 2;2(8):e199441. doi: 10.1001/jamanetworkopen.2019.9441. PMID 31418805